CLINICAL TRIAL: NCT04357379
Title: Impact Of IQOS Non-Cigarette Tobacco Product On Reinforcement Value and Use In Current Smokers
Brief Title: IQOS (Non-Cigarette Tobacco Product) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Tracy Smith, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00098672
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IQOS group (Experimental)
  Interventions: Behavioral: IQOS

INTERVENTIONS:
Behavioral: IQOS — Participants will try an IQOS product and then take home the IQOS to sample for one week.
  Other Names: heated tobacco product (HTP)

SUMMARY:
A novel type of non-cigarette tobacco product was recently approved for sale in the US, the heated tobacco product (HTP) IQOS. IQOS may be less harmful than cigarettes, and there are some reports that it may produce more rewarding subjective effects compared to e-cigarettes. The approval of IQOS provides a unique opportunity to gather preliminary data surrounding IQOS. The goal of this pilot study is to assess the subjective effects and relative reinforcement value of IQOS, including its downstream effects on cigarette smoking. Current smokers will complete a one-week baseline period where they smoke as normal before attending an in-person lab visit. During the in-person lab visit, participants (n=10) will sample a traditional cigarette and a novel IQOS tobacco product. Participants will answer questionnaires about each product they sample and then complete a preference assessment in which they choose between the IQOS and their own cigarette. Finally, participants will take home a tobacco product they sampled to use ad libitum (1-week sampling). During the at-home baseline and sampling weeks, participants will complete electronic daily diaries cataloging their tobacco use. Biomarkers (i.e., expired carbon monoxide, cotinine) will corroborate self-reported indices of use.

ELIGIBILITY:
Inclusion Criteria:

* daily cigarette smoker
* interested in using non-cigarette tobacco product
* have a smartphone that can receive text messages and has access to the internet or have an e-mail account they check daily (necessary for daily diary completion).

Exclusion Criteria:

* additional tobacco use criteria
* additional medical criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IQOS Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IQOS Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Prefer IQOS
Description: Participants complete a preference assessment in which they choose between the IQOS or a traditional cigarette in a series of trials. The outcome of this assessment is the number of participants who prefer the IQOS over a traditional cigarette
Time Frame: Lab Visit 2, occurring approximately one week after the initial screening/baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | IQOS Group
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Cigarettes Per Day
Description: The average percent reduction in cigarettes per day observed in Week 2
Time Frame: Week 2 of study
Measure: Mean (Standard Deviation); unit: Percentage reduction in cigs per day
Arm/Group | IQOS Group
Number analyzed (Participants) | 10
Percentage reduction in cigs per day | 16.1 (32.7)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Interviewer-administered assessment at each visit
Arm/Group | IQOS Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IQOS Group (N=10)
Cough (General disorders) | 1 (2)
Headache (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
ER visit for medication refill (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04357379/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT04357379/ICF_000.pdf